CLINICAL TRIAL: NCT06482749
Title: Impact of Repetitive Transcranial Magnetic Stimulation on Postoperative Neurocognitive Recovery in Older Patients With Preoperative Cognitive Impairment: A Randomized, Double-blinded, Sham-controlled Trial
Brief Title: Repetitive Transcranial Magnetic Stimulation and Postoperative Neurocognitive Recovery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Collaborators: The First Affiliated Hospital of Air Force Medicial University (Other); Peking University Shenzhen Hospital (Other)
Responsible Party: Principal Investigator, Dong-Xin Wang, Professor, Peking University First Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2024-232
Record Dates: First submitted 2024-06-23; First posted 2024-07-01 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Older Patients; Cognitive Impairment; Repetitive Transcranial Magnetic Stimulation; Delayed Neurocognitive Recovery; Postoperative Neurocognitive Disorder
Keywords: Older patients; Cognitive impairment; Repetitive transcranial magnetic stimulation; Delayed neurocognitive recovery; Postoperative neurocognitive disorder
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Repetitive Transcranial Magnetic Stimulation Group (Experimental): Repeated transcranial magnetic stimulation (rTMS) over left dorsolateral prefrontal cortex (DLPFC) for a 5-day period (1 day before surgery and 4 consecutive days after surgery, twice daily [10-12 am and 6-8 pm], no intervention on the day of the surgery). Parameters of rTMS: "8" shaped coil, 10 Hz, 80% resting motor threshold (RMT), 2000 pulses (5s × 40 trains, 25 s interval), 20 minutes.
  Interventions: Device: Repetitive transcranial magnetic stimulation
- Sham Stimulation Group (Sham Comparator): Sham repeated transcranial magnetic stimulation (rTMS) over left dorsolateral prefrontal cortex (DLPFC) for a 5-day period (1 day before surgery and 4 consecutive days after surgery, twice daily [10-12 am and 6-8 pm], no intervention on the day of the surgery). Parameters of rTMS: "8" shaped sham coil, 10 Hz, 80% resting motor threshold (RMT), 2000 pulses (5s × 40 trains, 25 s interval), 20 minutes.
  Interventions: Device: Sham stimulation

INTERVENTIONS:
Device: Repetitive transcranial magnetic stimulation — Repeated transcranial magnetic stimulation (rTMS) over left dorsolateral prefrontal cortex (DLPFC) for a 5-day period (1 day before surgery and 4 consecutive days after surgery, twice daily [10-12 am and 6-8 pm], no intervention on the day of the surgery). Parameters of rTMS: "8" shaped coil, 10 Hz, 80% resting motor threshold (RMT), 2000 pulses (5s × 40 trains, 25 s interval), 20 minutes.
  Arms: Repetitive Transcranial Magnetic Stimulation Group
Device: Sham stimulation — Sham repeated transcranial magnetic stimulation (rTMS) over left dorsolateral prefrontal cortex (DLPFC) for a 5-day period (1 day before surgery and 4 consecutive days after surgery, twice daily [10-12 am and 6-8 pm], no intervention on the day of the surgery). Parameters of rTMS: "8" shaped sham coil, 10 Hz, 80% resting motor threshold (RMT), 2000 pulses (5s × 40 trains, 25 s interval), 20 minutes.
  Arms: Sham Stimulation Group

SUMMARY:
Patients with preoperative cognitive impairment are at increased risks of delayed neurocognitive recovery (DNR) and postoperative neurocognitive disorder (POCD). Repetitive transcranial magnetic stimulation (rTMS) has been used to improve cognitive function in patients with cognitive impairement. This trial is designed to compare the effects of rTMS versus sham intervention on postoperative neurocognitive function in patients with preoperative cognitive impairment.

DETAILED DESCRIPTION:
Mild cognitive impairment (MCI) affects 10-15% of the population over 65 years old. In patients for elective non-cardiac and emergency surgeries, the pooled prevalences of unrecognized cognitive impairment were 37.0% and 50.0%, respectively. Patients with preoperative cognitive impairment are at increased risk of delayed neurocognitive recovery (DNR) and postoperative neurocognitive disorder (POCD). Therefore, perioperative neurocognitive protection is particularly important for patients with preoperative cognitive impairment.

Repetitive transcranial magnetic stimulation (rTMS) is a neural modulation technique. By acting on the brain and altering the membrane potential of cortical neurons, the generated pulsed magnetic fields affect neural metabolism and electrical activity and trigger a series of physiological and biochemical reactions. It was found that high frequency (>5 Hz) rTMS increases cortical excitability, whereas low frequency (<1Hz) rTMS reduces corticol excitability. The mechanism by which rTMS regulates brain function is generally believed to be related to the long-term enhancement and long-term inhibition of synaptic transmission function.

The left dorsolateral prefrontal cortex (DLPFC) is an important target of rTMS intervention for improving cognitive function. A meta-analysis showed that high-frequency rTMS on the DLPFC and low-frequency rTMS on the right medial prefrontal cortex improved memory function; high frequency rTMS on the right inferior frontal gyrus enhanced executive ability in non-surgical patients with mild cognitive impairment or Alzheimer's disease. Another meta-analysis showed that high-frequency rTMS on DLPFC is an effective therapeutic option for improving cognitive function in Alzheimer patients.

This trial is designed to compare the effects of rTMS versus sham intervention on postoperative neurocognitive function in patients with preoperative cognitive impairment.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥65 years;
2. Patients with preoperative mild to moderate cognitive impairment, defined as 9<Montreal Cognitive Assessment (MoCA)<26;
3. Scheduled for elective non-cardiac surgery under general anesthesia, with an expected surgical duration of >2 hours;
4. Expected to stay in hospital for at least 5 days after surgery.

Exclusion Criteria:

1. Left-handed;
2. Primary school education level or below;
3. Comorbid diseases including mental illness, intellectual disability, auditory and visual dysfunction, language impairment, severe neurological disorders, or other diseases that impede the completion of evaluation;
4. Neurosurgery;
5. Presence of contraindications to rTMS treatment, including epilepsy, pregnant or lactating women, or with a metal or electric implanted device (e.g., deep brain stimulator, ventriculoperitoneal shunt, aneurysm clip, pacemaker, cochlear implant, or surgical staples on the scalp);
6. Other situations that are deemed unsuitable for inclusion in the study.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 568 (Estimated)
Dates: Start 2025-07-28 (Actual); Primary Completion 2028-08 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Incidence of delayed neurocognitive recovery | On the 5th day after surgery
  Cognitive function is assessed with the Montreal Cognitive Assessment (MoCA; scores range from 0 to 30, with higher score indicating better function) before surgery and at 5 days after surgery. A MoCA score reduction of 1 standard deviation (SD) or more from baseline is defined as occurrence of delayed neurocognitive recovery.

SECONDARY OUTCOMES:
Incidence of delirium | Within 5 days after surgery
  Delirium is assessed with the 3D-Confusion Assessment Method (for non-intubated patients) or Confusion Assessment Method for the Intensive Care Unit (for intubated patients) twice daily (8-10 am and 4-6 pm).
Incidence of postoperative neurocognitive disorder at 30 days after surgery | On the 30(±3)th day after surgery
  Cognitive function is assessed with the Telephone Montreal Cognitive Assessment (T-MoCA; scores range from 0 to 22, with higher score indicating better function) at 30±3 days after surgery. A T-MoCA score reduction of 1 standard deviation (SD) or more from baseline is defined as occurrence of postoperative neurocognitive disorder.
Incidence of postoperative neurocognitive disorder at 180 days after surgery | On the 180(±15)th day after surgery
  Cognitive function is assessed with the Telephone Montreal Cognitive Assessment (T-MoCA; scores range from 0 to 22, with higher score indicating better function) at 180±15 days after surgery. A T-MoCA score reduction of 1 standard deviation (SD) or more from baseline is defined as occurrence of postoperative neurocognitive disorder.

OTHER OUTCOMES:
Pain intensity within 5 days after surgery | Up to 5 days after surgery
  Pain intnsity is assessed with the Numerical Rating Scale (NRS, an 11-point scale where 0 = no pain and 10 = the worst pain) twice daily (8-10 am and 4-6 pm) during the first 5 days after surgery.
Length hospital stay after surgery | Up to 30 days after surgery
  Length hospital stay after surgery.
Incidences of complications within 30 days after surgery | Up 30 days after surgery
  Postoperative complications are defined as new-onset medical events other than delirium that are deemed harmful and require therapeutic intervention, that is grade II or higher on the Clavien-Dindo classification.
Quality of life at 30 days after surgery | On the 30(±3)th day after surgery
  Quality of life is assessed with the World Health Organization Quality of Life brief version (WHOQOL-BREF), a 24-item questionnaire that assesses the quality of life in physical, psychological, and social relationship, and environmental domains. The score ranges from 0 to 100 for each domain, with higher score indicating better function.
Quality of life at 180 days after surgery | On the 180(±15)th day after surgery
  Quality of life is assessed with the World Health Organization Quality of Life brief version (WHOQOL-BREF), a 24-item questionnaire that assesses the quality of life in physical, psychological, and social relationship, and environmental domains. The score ranges from 0 to 100 for each domain, with higher score indicating better function.
Event-free survival within 180 days after surgery | Up to 180 days after surgery
  Time interval from index surgery to cancer recurrence/metastasis/progression, new-onset cancer, new-onset serious illness (requiring hospitalization), or all-cause death, whichever comes first.

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Xin Wang, MD, PhD, Principal Investigator — Peking University First Hospital
Locations (3):
- China (3):
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Peking University Shenzhen Hospital, Shenzhen, Guangzhou
  - Xijing Hospital, Air Force Medical University, Xi'an, Shannxi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Anderson ND. State of the science on mild cognitive impairment (MCI). CNS Spectr. 2019 Feb;24(1):78-87. doi: 10.1017/S1092852918001347. Epub 2019 Jan 17. PMID 30651152
- [Background] Kapoor P, Chen L, Saripella A, Waseem R, Nagappa M, Wong J, Riazi S, Gold D, Tang-Wai DF, Suen C, Englesakis M, Norman R, Sinha SK, Chung F. Prevalence of preoperative cognitive impairment in older surgical patients.: A systematic review and meta-analysis. J Clin Anesth. 2022 Feb;76:110574. doi: 10.1016/j.jclinane.2021.110574. Epub 2021 Nov 5. PMID 34749047
- [Background] Park S, Kim J, Ha Y, Kim KN, Yi S, Koo BN. Preoperative mild cognitive impairment as a risk factor of postoperative cognitive dysfunction in elderly patients undergoing spine surgery. Front Aging Neurosci. 2024 Jan 12;16:1292942. doi: 10.3389/fnagi.2024.1292942. eCollection 2024. PMID 38282693
- [Background] Silbert B, Evered L, Scott DA, McMahon S, Choong P, Ames D, Maruff P, Jamrozik K. Preexisting cognitive impairment is associated with postoperative cognitive dysfunction after hip joint replacement surgery. Anesthesiology. 2015 Jun;122(6):1224-34. doi: 10.1097/ALN.0000000000000671. PMID 25859906
- [Background] Hallett M. Transcranial magnetic stimulation: a primer. Neuron. 2007 Jul 19;55(2):187-99. doi: 10.1016/j.neuron.2007.06.026. PMID 17640522
- [Background] Du J, Yang F, Hu J, Hu J, Xu Q, Cong N, Zhang Q, Liu L, Mantini D, Zhang Z, Lu G, Liu X. Effects of high- and low-frequency repetitive transcranial magnetic stimulation on motor recovery in early stroke patients: Evidence from a randomized controlled trial with clinical, neurophysiological and functional imaging assessments. Neuroimage Clin. 2019;21:101620. doi: 10.1016/j.nicl.2018.101620. Epub 2018 Dec 3. PMID 30527907
- [Background] Wang Q, Zhang D, Zhao YY, Hai H, Ma YW. Effects of high-frequency repetitive transcranial magnetic stimulation over the contralesional motor cortex on motor recovery in severe hemiplegic stroke: A randomized clinical trial. Brain Stimul. 2020 Jul-Aug;13(4):979-986. doi: 10.1016/j.brs.2020.03.020. Epub 2020 Apr 2. PMID 32380449
- [Background] Chen Q, Shen W, Sun H, Zhang H, Liu C, Chen Z, Yu L, Cai X, Ke J, Li L, Zhang L, Fang Q. The effect of coupled inhibitory-facilitatory repetitive transcranial magnetic stimulation on shaping early reorganization of the motor network after stroke. Brain Res. 2022 Sep 1;1790:147959. doi: 10.1016/j.brainres.2022.147959. Epub 2022 May 30. PMID 35654120
- [Background] Gaudeau-Bosma C, Moulier V, Allard AC, Sidhoumi D, Bouaziz N, Braha S, Volle E, Januel D. Effect of two weeks of rTMS on brain activity in healthy subjects during an n-back task: a randomized double blind study. Brain Stimul. 2013 Jul;6(4):569-75. doi: 10.1016/j.brs.2012.10.009. Epub 2012 Nov 19. PMID 23194830
- [Background] Alcala-Lozano R, Morelos-Santana E, Cortes-Sotres JF, Garza-Villarreal EA, Sosa-Ortiz AL, Gonzalez-Olvera JJ. Similar clinical improvement and maintenance after rTMS at 5 Hz using a simple vs. complex protocol in Alzheimer's disease. Brain Stimul. 2018 May-Jun;11(3):625-627. doi: 10.1016/j.brs.2017.12.011. Epub 2017 Dec 29. PMID 29326021
- [Background] Bressler SL, Menon V. Large-scale brain networks in cognition: emerging methods and principles. Trends Cogn Sci. 2010 Jun;14(6):277-90. doi: 10.1016/j.tics.2010.04.004. Epub 2010 May 20. PMID 20493761
- [Background] Li Y, Wang L, Jia M, Guo J, Wang H, Wang M. The effects of high-frequency rTMS over the left DLPFC on cognitive control in young healthy participants. PLoS One. 2017 Jun 14;12(6):e0179430. doi: 10.1371/journal.pone.0179430. eCollection 2017. PMID 28614399
- [Background] Chou YH, Ton That V, Sundman M. A systematic review and meta-analysis of rTMS effects on cognitive enhancement in mild cognitive impairment and Alzheimer's disease. Neurobiol Aging. 2020 Feb;86:1-10. doi: 10.1016/j.neurobiolaging.2019.08.020. Epub 2019 Aug 27. PMID 31783330
- [Background] Simko P, Kent JA, Rektorova I. Is non-invasive brain stimulation effective for cognitive enhancement in Alzheimer's disease? An updated meta-analysis. Clin Neurophysiol. 2022 Dec;144:23-40. doi: 10.1016/j.clinph.2022.09.010. Epub 2022 Sep 28. PMID 36215904
- [Background] Gao Y, Qiu Y, Yang Q, Tang S, Gong J, Fan H, Wu Y, Lu X. Repetitive transcranial magnetic stimulation combined with cognitive training for cognitive function and activities of daily living in patients with post-stroke cognitive impairment: A systematic review and meta-analysis. Ageing Res Rev. 2023 Jun;87:101919. doi: 10.1016/j.arr.2023.101919. Epub 2023 Mar 31. PMID 37004840
- [Background] Chu CS, Li CT, Brunoni AR, Yang FC, Tseng PT, Tu YK, Stubbs B, Carvalho AF, Thompson T, Rajji TK, Yeh TC, Tsai CK, Chen TY, Li DJ, Hsu CW, Wu YC, Yu CL, Liang CS. Cognitive effects and acceptability of non-invasive brain stimulation on Alzheimer's disease and mild cognitive impairment: a component network meta-analysis. J Neurol Neurosurg Psychiatry. 2021 Feb;92(2):195-203. doi: 10.1136/jnnp-2020-323870. Epub 2020 Oct 28. PMID 33115936
- [Background] Miller A, Allen RJ, Juma AA, Chowdhury R, Burke MR. Does repetitive transcranial magnetic stimulation improve cognitive function in age-related neurodegenerative diseases? A systematic review and meta-analysis. Int J Geriatr Psychiatry. 2023 Aug;38(8):e5974. doi: 10.1002/gps.5974. PMID 37526325
- [Background] Zhang Y, Shan GJ, Zhang YX, Cao SJ, Zhu SN, Li HJ, Ma D, Wang DX; First Study of Perioperative Organ Protection (SPOP1) investigators. Propofol compared with sevoflurane general anaesthesia is associated with decreased delayed neurocognitive recovery in older adults. Br J Anaesth. 2018 Sep;121(3):595-604. doi: 10.1016/j.bja.2018.05.059. Epub 2018 Jul 27. PMID 30115258
- [Background] Jeste DV, Palmer BW, Appelbaum PS, Golshan S, Glorioso D, Dunn LB, Kim K, Meeks T, Kraemer HC. A new brief instrument for assessing decisional capacity for clinical research. Arch Gen Psychiatry. 2007 Aug;64(8):966-74. doi: 10.1001/archpsyc.64.8.966. PMID 17679641